CLINICAL TRIAL: NCT04273217
Title: A Phase 1a, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Determine the Safety and Pharmacokinetics of AV-1 in Healthy Male and Female Adult Subjects
Brief Title: A Study to Determine the Safety of AV-1, an Antibody Being Developed for Treatment of Dengue, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbViro LLC (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: AV1-PPD-0005; DMID 18-0016 (Other: DMID Protocol Number); HHSN272201600028C (Other: NIAID Contract Number)
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Monoclonal antibody; AV-1; Safety; Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- AV-1 30 mg (Experimental): Participants received a single intravenous (IV) infusion (infusion duration: 1 hour) of AV-1 30 mg on Day 1.
  Interventions: Drug: AV-1
- AV-1 90 mg (Experimental): Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 90 mg on Day 1.
  Interventions: Drug: AV-1
- AV-1 250 mg (Experimental): Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 250 mg on Day 1.
  Interventions: Drug: AV-1
- AV-1 500 mg (Experimental): Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 500 mg on Day 1.
  Interventions: Drug: AV-1
- AV-1 1000 mg (Experimental): Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 1000 mg on Day 1.
  Interventions: Drug: AV-1
- Placebo (Placebo Comparator): Participants received a single IV infusion (infusion duration: 1 hour) of placebo matched to AV-1 on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AV-1 — Single dose, administered by IV infusion (volume: 250 mL)
  Arms: AV-1 1000 mg; AV-1 250 mg; AV-1 30 mg; AV-1 500 mg; AV-1 90 mg
Drug: Placebo — 0.9% sterile saline. Administered by IV infusion (volume: 250 mL)
  Arms: Placebo

SUMMARY:
AV-1 is a human monoclonal antibody (mAb) being investigated as a potential therapy for dengue, a mosquito-borne viral disease with extensive global public health impact. Globally, over 2 billion people are thought to be at risk of infection from the dengue virus and there are an estimated 390 million infections each year. Current treatment options for dengue are limited to supportive care, so a safe and effective treatment would provide substantial public health benefits. AV-1 has not previously been tested in humans. This study aims to determine the safety of AV-1 in healthy adult volunteers, when administered as a single IV infusion. The results of the study are based on the clinical study report and statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be in good health at Screening (reaffirmed at Check-in):

  1. Good health is defined by the absence of a medical condition described in the exclusion criteria of the study protocol, and based on screening medical history, physical examination, vital signs, and 12-lead electrocardiogram (ECG).
  2. If the subject has another current, ongoing chronic medical condition, the condition cannot: (i) Be first diagnosed within 3 months of enrollment; or (ii) Be a pre-existing medical condition that is not exclusionary but has worsened in terms of clinical outcome within 3 months of enrollment; or (iii) Involve the need for medication that may pose a risk to the subject's safety or impede assessment of adverse events (AEs) or anti-AV-1 antibody response if they participate in the study.
* Women who are not pregnant and/or not lactating.
* Female subjects, including postmenopausal women and surgically sterile women, must have a negative serum pregnancy test at Screening, Check-in and on admission to the study facility.
* Female subjects must fulfill one of the following criteria:

  1. Postmenopausal women must have had ≥ 12 months of spontaneous amenorrhea with follicle-stimulating hormone concentration consistently ≥40 mIU/mL and must have a negative pregnancy test result at Screening and Check-in.
  2. Surgically sterile women - those who have had a hysterectomy, bilateral ovariectomy (oophorectomy), or bilateral tubal ligation, must provide documentation of the procedure and must have a negative pregnancy test at Screening and Check-in.
  3. Must be willing to not engage in sexual intercourse from Check-in until the final follow-up visit on Day 120 (± 5 days).
  4. Must be willing to use an acceptable method of birth control until the final follow-up visit on Day 120 (± 5 days) as defined by the protocol and Investigator.
* Male subjects who are biologically capable of fathering children must agree and commit to using an adequate form of double-barrier contraception, and refrain from sperm donation from Check-in until the final follow-up visit on Day 120 (± 5 days). A male subject is considered capable of fathering children even if his sexual partner is sterile or using contraceptives.
* Body Mass Index between 18.5 and 29.9 kg/m^2 inclusive.
* Must not have traveled outside the USA within 60 days prior to Check-in, and agree not to travel outside the USA through the final follow-up visit on Day 120 (± 5 days).
* Must agree to abide by study restrictions and be willing to sign an informed consent form (ICF).

Exclusion Criteria:

* Any significant medical condition that, in the opinion of the Investigator or Sponsor, would interfere with the subject's ability to participate in the study or increase the risk of participating for that subject, based on the Investigator's Brochure and the safety profile of AV-1.
* Subject has one or more symptoms of a urinary tract infection (e.g. dysuria, frequent, urgency, or suprapubic pain) at Screening or Check-in.
* Has certain abnormal12-lead ECG (electrocardiogram) results according to the protocol, as assessed by the Investigator.
* Has abnormal laboratory values for certain hematology, serum chemistry, coagulation, or urinalysis tests according to the protocol, as assessed by the Investigator.
* Is positive for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody types 1 and 2 within 35 days of enrollment.
* Has any psychiatric condition or history of psychiatric condition that, in the opinion of the Investigator or Sponsor, would interfere with the subject's ability to participate in the study or increase the risk of participation for that subject.
* Is unwilling to abstain from alcohol, caffeine-, or other xanthine-containing foods or beverages, tobacco or nicotine-containing products, and all bergamottin-containing fruits and fruit juices (e.g. Seville oranges, grapefruit/grapefruit juice, pomelos, pomegranate/pomegranate juice, cranberries/cranberry juice) 72 hours prior to Check-in, through discharge on Day 5 of the study.
* Is unwilling to abstain from strenuous exercise 7 days before Check-in through Day 15 of the study.
* Has a history of alcoholism or drug/chemical abuse within 6 months prior to Check-in.
* Has excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects) (1 unit is equal to approximately 1/2 pint [200 mL] beer, 1 small glass [100 mL] wine, or 1 measure [25 mL] spirits).
* Has a positive urine drug screen at Screening or Check-in.
* Has a positive cotinine urine test at Check-in.
* Has any confirmed or suspected immunosuppressive or immunodeficient condition, including but not limited to human immunodeficiency virus infection, or use of anti-cancer chemotherapy or radiation therapy (cytotoxic) in the 3 years prior to Screening.
* Provides verbal history of vaccination with a licensed or investigational flavivirus vaccine for any of the following diseases: Zika virus, dengue virus (DENV), yellow fever virus, Japanese encephalitis virus, West Nile virus, St. Louis encephalitis virus, or tick-borne encephalitis virus; or reportedly diagnosed with a flavivirus infection or disease.
* Plans to receive a licensed flavivirus vaccine or participate in flavivirus vaccine trial during the study.
* Is positive for DENV or West Nile virus by immunoglobulin M, or immunoglobulin G, or Zika by immunoglobulin M serology testing within 35 days of enrollment.
* Has a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* Has had major surgery within 3 months prior to Screening or plans to have major surgery during the study through the final follow-up on Day 120 (± 5 days).
* Has been treated for a medical condition with a licensed monoclonal or polyclonal antibody in the past; or dosed in a clinical study involving administration of an investigational monoclonal or polyclonal antibody in the 18 months prior to study drug administration on Day 1.
* Has received an investigational drug within 28 days of study drug administration on Day 1.
* Has used any prohibited medication within 30 days prior to Check-in, or plans to use prohibited medication during the study. Prohibited medications include: Immunosuppressive drugs, immune modulators (except acetaminophen), oral corticosteroids, inhaled or intranasal steroids (<800 µg/day beclomethasone is acceptable), and anti-neoplastic agents. Topical steroids are acceptable.
* Has received or plans to receive any live vaccination, experimental or otherwise, within 28 days prior to or after Day 1 of the study; and receipt or planned receipt of an inactivated vaccination (or any COVID-19 vaccine), experimental or otherwise, within 14 days prior to or after Day 1 of the study.
* Has received blood products within 60 days prior to Check-in.
* Has donated or lost more than 450 mL of blood or plasma within 56 days of study drug infusion on Day 1. The subject must also agree to refrain from donating blood or plasma during the study.
* Has poor peripheral venous access.
* Previously completed or withdrawn from this study.
* Is a current clinical site staff paid entirely or partially by the contractor for this trial, or staff who are supervised by the Investigator or subinvestigators.
* In the opinion of the Investigator (or designee), the subject is not suitable for entry into the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wood-Horrall, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Austin Clinic, 7551 Metro Center Drive, Suite 200, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Medical Product Safety Information — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: FDA Recalls, Market Withdrawals, and Safety Alerts — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center study conducted in the United States.
Pre-assignment Details: On the first day of dosing in all cohorts, the first group in each cohort comprised 2 sentinel participants: 1 was randomly assigned to receive AV-1 and the other was randomly assigned to receive placebo. After the Investigator reviewed the safety data from the 72-hour post-dose period for the sentinel participants, the remainder of the cohort (5 participants randomly assigned to AV-1; 1 participant randomly assigned to placebo) were dosed at least 72 hours after the sentinel participants.
Groups:
- AV-1 30 mg: Participants received a single intravenous (IV) infusion (infusion duration: 1 hour) of AV-1 30 mg (volume: 250 mL) on Day 1.
- AV-1 90 mg: Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 90 mg (volume: 250 mL) on Day 1.
- AV-1 250 mg: Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 250 mg (volume: 250 mL) on Day 1.
- AV-1 500 mg: Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 500 mg (volume: 250 mL) on Day 1.
- AV-1 1000 mg: Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 1000 mg (volume: 250 mL) on Day 1.
- Placebo: Participants received a single IV infusion (infusion duration: 1 hour) of placebo (volume: 250 mL) on Day 1.
Period: Overall Study
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Started | 6 | 6 | 6 | 6 | 7 | 11
Completed | 5 | 6 | 5 | 6 | 6 | 9
Not Completed | 1 | 0 | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant non-compliance | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Positive urine drug screen | 1 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety population included all participants who received any amount of the investigational product.
Groups:
- AV-1 30 mg: Participants received a single IV infusion (infusion duration: 1 hour) of AV-1 30 mg (volume: 250 mL) on Day 1.
- Total: Total of all reporting groups
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (6.89) | 35.0 (9.65) | 35.0 (9.72) | 32.3 (8.29) | 37.0 (13.52) | 35.4 (10.50) | 36.4 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 3 | 4 | 4 | 6 | 25
  Male | 0 | 4 | 3 | 2 | 3 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 4 | 3 | 5 | 17
  Not Hispanic or Latino | 3 | 5 | 5 | 2 | 4 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 0 | 1 | 1 | 3 | 7
  White | 4 | 3 | 5 | 5 | 6 | 8 | 31
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Clinical laboratory abnormalities reported as TEAEs by the investigator. Clinical laboratory abnormalities were defined as any abnormal findings in analysis of hematology, serum chemistry, coagulation, and urine parameters. A TEAE was defined as any event not present before exposure to study drug or any event already present that worsened in intensity or frequency after exposure whether or not considered drug related.
Time Frame: Baseline up to Day 120 (± 5 days)
Population: The Safety population included all participants who received any amount of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11
Participants
  Hematology (blood glucose increased) | 0 | 0 | 0 | 0 | 1 | 0
  Serum chemistry | 0 | 0 | 0 | 0 | 0 | 0
  Coagulation | 0 | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Physical Examination Abnormalities Reported as TEAEs
Description: A full physical examination included examination of skin; head, ears, eyes, nose, throat (HEENT); neck; thyroid; lungs; heart; cardiovascular; abdomen; lymph nodes; and musculoskeletal system/extremities. Focused examination included lungs, cardiovascular, abdomen, and skin. Investigator could perform targeted, symptom-directed physical examination. A TEAE was defined as any event not present before exposure to study drug or any event already present that worsened in intensity or frequency after exposure whether or not considered drug related.
Time Frame: Baseline up to Day 120 (± 5 days)
Population: Participants in the Safety Population were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11
Participants
  Abdomen | 0 | 0 | 0 | 0 | 0 | 0
  Cardiovascular | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal system/extremities | 0 | 0 | 0 | 0 | 0 | 0
  Heart | 0 | 0 | 0 | 0 | 0 | 0
  HEENT | 0 | 0 | 0 | 0 | 0 | 0
  Lungs | 0 | 0 | 0 | 0 | 0 | 0
  Lymph nodes | 0 | 0 | 0 | 0 | 0 | 0
  Neck | 0 | 0 | 0 | 0 | 0 | 0
  Skin (dermatitis contact) | 0 | 0 | 0 | 0 | 1 | 0
  Thyroid | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Vital Sign Abnormalities Reported as TEAEs
Description: Vital sign measurements included systolic and diastolic blood pressure, oral body temperature, heart rate, and respiratory rate. A TEAE was defined as any event not present before exposure to study drug or any event already present that worsened in intensity or frequency after exposure whether or not considered drug related.
Time Frame: Baseline up to Day 120 (± 5 days)
Population: Participants in the Safety Population were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With 12-lead Electrocardiogram (ECG) Abnormalities Reported as TEAEs
Description: Number of participants with abnormal 12-lead ECG reported as a TEAE of electrocardiogram QT prolonged by the investigator. A TEAE was defined as any event not present before exposure to study drug or any event already present that worsened in intensity or frequency after exposure whether or not considered drug related.
Time Frame: Baseline up to Day 120 (± 5 days)
Population: Participants in the Safety Population were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11
Participants | 2 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Number of Participants With TEAEs
Description: An adverse event (AE) was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. A TEAE was defined as any event not present before exposure to study drug or any event already present that worsened in intensity or frequency after exposure.
Time Frame: Baseline up to Day 120 (± 5 days)
Population: Participants in the Safety Population were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11
Participants | 3 | 3 | 0 | 1 | 4 | 3

6. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE or suspected adverse reaction was considered an SAE if, in the view of either the Investigator or Sponsor, it resulted in any of the following outcome:
  * Death
  * A life-threatening AE
  * Inpatient hospitalization or prolongation of existing hospitalization
  * a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital anomaly/birth defect
  Important medical events that did not result in death, was life-threatening, or required hospitalizations could have been considered serious when, based upon appropriate medical judgment, they jeopardized the participant and required medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Baseline up to Day 120 (± 5 days)
Population: Participants in the Safety Population were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants by Severity of AEs
Description: AEs were assessed by the Investigator as Mild (Grade 1), Moderate (Grade 2), or Severe (Grade 3).
  Mild (Grade 1): Events that were transient and required only minimal or no treatment or therapeutic intervention and did not interfere with the participants usual activities of daily living.
  Moderate (Grade 2): Events that were alleviated with additional specific therapeutic intervention. The event interfered with usual activities of daily living, causing discomfort but posed no significant or permanent risk of harm to the participant.
  Severe (Grade 3): Events interrupted usual activities of daily living, or significantly affected clinical status, or required intensive therapeutic intervention. Severe events were usually incapacitating.
Time Frame: Baseline up to Day 120 (± 5 days)
Population: Participants in the Safety Population who experienced any AE were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 3 | 3 | 0 | 1 | 4 | 3
Participants
  Mild | 1 | 3 | 0 | 1 | 3 | 3
  Moderate | 2 | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 1 | 0

8. Secondary Outcome: Area Under the Serum Concentration-time Curve (AUC) From Time 0 Extrapolated to Infinity (AUC0-infinity) of AV-1
Description: AUC0-infinity was calculated as: AUC from time 0 to the last quantifiable concentration (AUC0-tlast) + (last observed serum drug concentration [Ct] / Apparent terminal elimination rate constant [λz]).
Time Frame: Predose (within 15 minutes); at 0.5, 1 (end of infusion), 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours after the start of infusion; Days 5, 8, 15, 22, 29, 43, 57, 85, and 120
Population: The pharmacokinetic (PK) population included participants who received the full dose of AV-1 and had at minimum all samples from predose through 1.5 hours from the start of infusion and had sufficient concentration data to support accurate estimation of at least 1 PK parameter. As placebo group did not receive AV-1, PK analysis for placebo group is not applicable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hour/mL
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
μg*hour/mL | 7940 (14.9) | 16700 (29.7) | 52800 (33.7) | 136000 (48.1) | 250000 (15.8)

9. Secondary Outcome: AUC From Time 0 to 48 Hours Postdose (AUC0-48) of AV-1
Description: AUC0-48 was calculated using the linear trapezoidal rule method.
Time Frame: Predose (within 15 minutes); at 0.5, 1 (end of infusion), 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, and 48 hours after the start of infusion
Population: Participants in the PK Population who have were analyzed. As placebo group did not receive AV-1, PK analysis for placebo group is not applicable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hour/mL
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
μg*hour/mL | 443 (16.1) | 1340 (19.7) | 3380 (20.7) | 11400 (74.1) | 16000 (20.2)

10. Secondary Outcome: AUC From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast)
Description: AUC0-tlast was calculated using the linear trapezoidal method.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hour/mL
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
μg*hour/mL | 7140 (12.4) | 15900 (27.9) | 48300 (30.6) | 129000 (48.0) | 233000 (16.7)

11. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of AV-1
Description: Cmax is defined as maximum observed serum drug concentration.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
μg/mL | 12.7 (10.8) | 41.8 (13.6) | 98.0 (22.0) | 332 (72.0) | 654 (87.2)

12. Secondary Outcome: Time to Reach Cmax (Tmax) of AV-1
Description: Tmax is defined as Time to reach maximum serum concentration following drug administration.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
hours | 2.00 [1.57 to 12.00] | 4.00 [1.00 to 8.00] | 1.38 [1.00 to 3.00] | 2.49 [1.00 to 4.00] | 2.00 [1.00 to 6.05]

13. Secondary Outcome: Apparent Terminal Half-life (t1/2) of AV-1
Description: t1/2 is defined as terminal half-life, calculated as: ln(2)/ λz, where λz is apparent terminal elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
hours | 910 (15.8) | 631 (25.0) | 768 (33.8) | 700 (24.4) | 732 (19.5)

14. Secondary Outcome: Total Serum Clearance (CL) of AV-1
Description: Total serum clearance was calculated as dose divided by AUC0-infinity.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
Liter/hour | 0.00378 (14.9) | 0.00539 (29.7) | 0.00474 (33.7) | 0.00366 (48.1) | 0.00399 (15.8)

15. Secondary Outcome: Volume of Distribution During the Terminal Phase (Vz) of AV-1
Description: Volume of distribution during the terminal phase was calculated as dose divided by (AUC0-infinity*λz).
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
Liter | 4.96 (9.0) | 4.90 (21.7) | 5.25 (24.0) | 3.70 (53.6) | 4.22 (25.0)

16. Secondary Outcome: Number of Participants With Detectable Anti-AV-1 Antibody
Description: Serum samples for measurement of anti-AV-1 antibody levels were analyzed by a validated electrochemiluminescence enzyme-linked immunosorbent assay method used for detection and confirmation of pre-existing and treatment-emergent anti-AV-1 antibodies in serum samples based on the MesoScale Discovery platform that utilized labeled AV-1 for detection of anti-AV-1 antibodies and treatment-emergent antibodies. Number of participants with detectable anti-AV-1 antibody
Time Frame: Baseline, Days 29 (±2), 85 (±5), and 120 (±5)
Population: Participants in the Safety Population were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 11
Participants
  Baseline | 0 | 0 | 1 | 0 | 0 | 0
  Day 29 (±2) | 0 | 0 | 0 | 0 | 0 | 0
  Day 85 (±5) | 0 | 0 | 0 | 0 | 0 | 0
  Day 120 (±5) | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 120 (± 5 days)
Description: The Safety population included all participants who received any amount of the investigational product.
Arm/Group | AV-1 30 mg | AV-1 90 mg | AV-1 250 mg | AV-1 500 mg | AV-1 1000 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/11
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 0/6 | 1/6 | 4/7 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AV-1 30 mg (N=6) | AV-1 90 mg (N=6) | AV-1 250 mg (N=6) | AV-1 500 mg (N=6) | AV-1 1000 mg (N=7) | Placebo (N=11)
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT04273217/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT04273217/SAP_001.pdf